CLINICAL TRIAL: NCT00613795
Title: Lactobacillus GG in the Prophylaxis of Ventilator Associated Pneumonia: A Prospective, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Lactobacillus GG in the Prophylaxis of Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Lee Morrow, MD, Creighton University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 03-13013
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Pneumonia; Ventilator Associated Pneumonia
Keywords: pneumonia; ventilator associated pneumonia; probiotics; Lactobacillus GG
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lactobacillus
  Interventions: Dietary Supplement: Lactobacillus GG
- 2 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG — Every 12 hours, the contents of a single capsule containing Lactobacillus GG will be suspended in 3 ml of water-soluble jelly. The suspension will be applied to the oropharyngeal mucosa via sterile syringe. The contents of a second capsule will be suspended in 10 ml of sterile water and pushed through the NG tub followed by 10 mL of air to ensure complete administration.
  Arms: 1
Dietary Supplement: placebo — Every 12 hours, the contents of a single identical placebo capsule containing the inert plant carbohydrate inulin will be suspended in 3 ml of water-soluble jelly. This suspension will be applied to the oropharyngeal mucosa via sterile syringe. The contents of a second placebo capsule will be suspended in 10 ml of sterile water and pushed through eh NG tube followed by 10 mL of air to ensure complete administration
  Arms: 2

SUMMARY:
This study utilizes lactobacillus, or probiotics, delivered twice daily to the mouth and stomach, via feeding tube, in effort to determine whether the oral administration of a naturally occurring Lactobacillus species reduces the incidence of ventilator associated pneumonia therefore reducing intensive care unit(ICU)complications.

DETAILED DESCRIPTION:
The long-term objective of this research is to determine the utility of altering the oral and gastric bacterial flora in mechanically ventilated patients in order to reduce intensive care unit (ICU)complications. Specifically, our goal is to determine whether the oral administration of a naturally occurring Lactobacillus species reduces the incidence of ventilator associated pneumonia (VAP). ICU admission is commonly accompanied by overgrowth of the natural gastrointestinal (GI) and oropharyngeal flor by pathogenic organisms. Patients requiring endotracheal intubation are predisposed to developing VAP, presumably via micro-aspiration of the altered oropharyngeal flora. By reducing VAP rates, we hope to improve ICU outcomes, minimize ICU expenses, and most importantly, decrease morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the medical, surgical, or cardiac ICU
* Age 19 years or greater (the age of majority in the state of Nebraska)
* Anticipated need for >72 hours of endotracheal intubation
* Initial intubation during hospitalization
* Approval of the attending physician responsible for the patient's care
* Informed surrogate consent within 24 hours of intubation

Exclusion Criteria:

* Pregnancy
* Pharmacologic immunosuppression (>10mg prednisone daily or equivalent for at least 14 days)
* Native immunosuppression: 1)known HIV disease or AIDS, 2)history of malignancy, 3)multiple organ system failure
* History of prosthetic or bioprosthetic cardiac valve placement
* History of prosthetic vascular graft placement
* Cardiac trauma
* History of rheumatic fever, endocarditis, congenital cardia abnormality, or acquired cardia abnormality
* Gastroesophageal surgery or perforation associated with current admission
* Intestinal surgery or perforation associated with current admission
* Significant oropharyngeal mucosal injury
* Placement of a tracheostomy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2004-08; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine whether patients given oral Lactobacillus GG will have a smaller increase in the density of pathogenic bacterial in cultures from oral swabs, nasogastric aspirates, and minimally invasive bronchoalveolar lavage samples. | daily while intubated

SECONDARY OUTCOMES:
To assess whether administration of Lactobacillus GG to intubated patients reduces clinically diagnosed VAP,reduces microbiologically diagnosed VAP, affects mortality and duration of mechanical ventilation, and total antibiotic consumption. | daily while intubated

CONTACTS AND LOCATIONS:
Overall Officials: Lee Morrow, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Atherton ST, White DJ. Stomach as source of bacteria colonising respiratory tract during artificial ventilation. Lancet. 1978 Nov 4;2(8097):968-9. doi: 10.1016/s0140-6736(78)92530-8. PMID 81991
- [Background] Ben-Menachem T, Fogel R, Patel RV, Touchette M, Zarowitz BJ, Hadzijahic N, Divine G, Verter J, Bresalier RS. Prophylaxis for stress-related gastric hemorrhage in the medical intensive care unit. A randomized, controlled, single-blind study. Ann Intern Med. 1994 Oct 15;121(8):568-75. doi: 10.7326/0003-4819-121-8-199410150-00003. PMID 8085688
- [Background] Bengmark S, Gianotti L. Nutritional support to prevent and treat multiple organ failure. World J Surg. 1996 May;20(4):474-81. doi: 10.1007/s002689900075. PMID 8662138
- [Background] Craven DE, Steger KA, Barber TW. Preventing nosocomial pneumonia: state of the art and perspectives for the 1990s. Am J Med. 1991 Sep 16;91(3B):44S-53S. doi: 10.1016/0002-9343(91)90343-v. PMID 1928191
- [Background] Hatakka K, Savilahti E, Ponka A, Meurman JH, Poussa T, Nase L, Saxelin M, Korpela R. Effect of long term consumption of probiotic milk on infections in children attending day care centres: double blind, randomised trial. BMJ. 2001 Jun 2;322(7298):1327. doi: 10.1136/bmj.322.7298.1327. PMID 11387176
- [Background] Fagon JY, Chastre J, Hance AJ, Montravers P, Novara A, Gibert C. Nosocomial pneumonia in ventilated patients: a cohort study evaluating attributable mortality and hospital stay. Am J Med. 1993 Mar;94(3):281-8. doi: 10.1016/0002-9343(93)90060-3. PMID 8452152
- [Background] Holzapfel WH, Haberer P, Geisen R, Bjorkroth J, Schillinger U. Taxonomy and important features of probiotic microorganisms in food and nutrition. Am J Clin Nutr. 2001 Feb;73(2 Suppl):365S-373S. doi: 10.1093/ajcn/73.2.365s. PMID 11157343
- [Background] Isolauri E. Probiotics in human disease. Am J Clin Nutr. 2001 Jun;73(6):1142S-1146S. doi: 10.1093/ajcn/73.6.1142S. PMID 11393192
- [Background] Johanson WG, Pierce AK, Sanford JP. Changing pharyngeal bacterial flora of hospitalized patients. Emergence of gram-negative bacilli. N Engl J Med. 1969 Nov 20;281(21):1137-40. doi: 10.1056/NEJM196911202812101. No abstract available. PMID 4899868
- [Background] Johanson WG Jr, Pierce AK, Sanford JP, Thomas GD. Nosocomial respiratory infections with gram-negative bacilli. The significance of colonization of the respiratory tract. Ann Intern Med. 1972 Nov;77(5):701-6. doi: 10.7326/0003-4819-77-5-701. No abstract available. PMID 5081492
- [Background] Johanson WG Jr, Seidenfeld JJ, de los Santos R, Coalson JJ, Gomez P. Prevention of nosocomial pneumonia using topical and parenteral antimicrobial agents. Am Rev Respir Dis. 1988 Feb;137(2):265-72. doi: 10.1164/ajrccm/137.2.265. PMID 3341620
- [Background] Rayes N, Seehofer D, Hansen S, Boucsein K, Muller AR, Serke S, Bengmark S, Neuhaus P. Early enteral supply of lactobacillus and fiber versus selective bowel decontamination: a controlled trial in liver transplant recipients. Transplantation. 2002 Jul 15;74(1):123-7. doi: 10.1097/00007890-200207150-00021. PMID 12134110
- [Background] Saavedra JM. Clinical applications of probiotic agents. Am J Clin Nutr. 2001 Jun;73(6):1147S-1151S. doi: 10.1093/ajcn/73.6.1147S. PMID 11393193
- [Background] Vanderhoof JA. Probiotics: future directions. Am J Clin Nutr. 2001 Jun;73(6):1152S-1155S. doi: 10.1093/ajcn/73.6.1152S. PMID 11393194
- [Derived] Morrow LE, Kollef MH, Casale TB. Probiotic prophylaxis of ventilator-associated pneumonia: a blinded, randomized, controlled trial. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1058-64. doi: 10.1164/rccm.200912-1853OC. Epub 2010 Jun 3. PMID 20522788